CLINICAL TRIAL: NCT01585415
Title: A Pilot Trial of the Combination of Vemurafenib With Adoptive Cell Therapy in Patients With Metastatic Melanoma
Brief Title: Vemurafenib and White Blood Cell Therapy for Advanced Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120114; 12-C-0114
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2016-07-21

CONDITIONS: Metastatic Cancer; Melanoma
Keywords: Tumor Infiltrating Lymphocytes; Immunotherapy; Adoptive Cell Therapy; B Raf Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — Vemurafenib; Cyclophosphamide; fludarabine; aldesleukin

ARMS (1):
- Single Arm (Experimental): Two weeks prior to the start of the preparative regimen, patients will begin taking vemurafenib. Patients will then receive lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine, followed by young TIL and high dose aldesleukin
  Interventions: Drug: Vemurafenib; Biological: Young TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib will administered orally twice a day at a dose of 960 mg from day -21 (+/- 7 days)until disease progression or patients are taken off protocol.
Biological: Young TIL — Young TIL will be administered intravenously on day 0(1x10e9 to 2x10e11) in the Patient Care Unit over 20-30 minutes via non-filtered tubing, gently agitating the bag during infusion to prevent cell clumping.
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with Mesna 15 mg/kg/day X 2 days over 1 hr.
Drug: Fludarabine — Fludarabine 25 mg/m2/day IVPB daily over 30 minutes for 5 days.
Drug: Aldesleukin — Aldeskeukin 720,000 IU/kg IV (based on total body weight)over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses)

SUMMARY:
Background:

- One possible treatment for advanced melanoma involves collecting white blood cells from the person with cancer and growing them in a laboratory. The cells can then be given back to the donor. This study will use this white blood cell treatment with the cancer treatment drug vemurafenib. Vemurafenib targets melanoma cells that have a mutation in the B-raf gene, and may be able to make them shrink.

Objectives:

- To see if vemurafenib and white blood cell therapy is a safe and effective treatment for advanced melanoma.

Eligibility:

- Individuals at least 18 years and less than or equal to 66 years of age who have advanced melanoma that contains the B-raf genetic mutation.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* White blood cells will be collected from tumor cells. These cells will be collected during surgery or a tumor biopsy.
* Participants will have leukapheresis to collect additional white blood cells for the procedure.
* Participants will take vemurafenib twice a day, starting 3 weeks before receiving the white blood cells.
* Participants will have 1 week of chemotherapy to prepare their immune system to accept the white blood cells.
* Participants will receive an infusion of their collected white blood cells. They will also receive aldesleukin for up to 5 days to boost the immune system s response to the white blood cells. They will remain in the hospital until they have recovered from the treatment.
* Participants will have frequent follow-up visits to monitor the outcome of the treatment.

DETAILED DESCRIPTION:
Background:

Adoptive cell therapy (ACT) with tumor infiltrating lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered to the autologous patient along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen.

Vemurafenib (VEM) administration has been shown to mediate objective responses in 50-60 percent of patients with metastatic melanoma bearing a BRAF mutation though many of these responses are transient.

There are several reasons to suggest that the combination of ACT with VEM will synergize in the destruction of melanoma including 1) rapid tumor destruction by VEM may provide a vaccine-like stimulus to the transferred TIL; 2) VEM has been shown to upregulate the expression of melanoma antigens; 3)VEM may make residual melanoma cells more sensitive to immune damage.

Objectives:

The primary objective is to determine the safety of the administration of vemurafenib in conjunction with ACT consisting of autologous TIL infused along with high dose aldesleukin following a non-myeloablative lymphodepleting preparative regimen.

The secondary objectives are:

* To gain preliminary information concerning the ability of the combination therapy to mediate clinical tumor regression in patients with metastatic melanoma.
* To study the immunologic impact of VEM administration on the lymphoid infiltrate in melanoma deposits.

Eligibility:

Patients greater than or equal to 18 years old with pathologically confirmed diagnosis of

metastatic melanoma that expresses the VtoE BRAF mutation and VtoK BRAF mutation.

Patients with measurable disease, absolute neutrophil count greater than 1000/mm(3) and platelet count greater than 100,000/mm(3).

No serious comorbid conditions such as active systemic infections, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory or immune systems.

Design:

Patients will undergo biopsy or resection to obtain tumor for generation of autologous TIL cultures.

When cryopreserved TIL are available patients will begin the administration of VEM 960 mg (day 1) twice daily until disease progression or patients are taken off protocol.

On day -7, patients will begin a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m2/day IV) on days -5 through -1.

On day 0, patients will receive between 1x109 to 2x1011 young TIL and then begin high dose aldesleukin (720,000 IU/kg IV every 8 hours for up to 15 doses).

Clinical and immunologic responses will be evaluated about 4-6 weeks after the last dose of aldesleukin.

This pilot trial will accrue 25 patients.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma that expresses the VtoE BRAF mutation and VtoK BRAF mutation assessed in a CLIA certified laboratory.
2. Patients with 3 or less brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
3. Greater than or equal to 18 and less than or equal to 66 years of age.
4. Patients of both genders must be willing to practice birth control from the time of enrollment on the study and for four months after treatment.
5. Life expectancy of greater than three months
6. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
7. Willing to sign a durable power of attorney.
8. Able to understand and sign the Informed Consent Document
9. Clinical performance status of ECOG 0 or 1.
10. Hematology:

    * Absolute neutrophil count greater than 1000/mm(3)
    * Hemoglobin greater than 8.0 g/dl
    * Platelet count greater than 100,000/mm(3)
11. Serology:

    * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, or hepatitis C antibody or antigen.
12. Chemistry:

    * Serum ALT/AST less than three times the upper limit of normal.
    * Calculated creatinine clearance (eGFR) > 50 ml/min.
    * Total bilirubin less than or equal to 2 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3 mg/dl.
13. More than four weeks must have elapsed since any prior systemic therapy at the time of treatment, and patients toxicities must have recovered to a grade 1 or less (except for alopecia or vitiligo). Patients must have stable or progressing disease after prior treatment.

    Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
14. Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-CTLA4 antibody therapy at the time the patient receives the preparative regimen to allow antibody levels to decline.

    Note: Patients who have previously received ipilimumab and have documented GI toxicity must have a normal colonoscopy with normal colonic biopsies.
15. EKG with mean QTc interval < 450 msec.

EXCLUSION CRITERIA:

1. Prior cell transfer therapy which included a myeloablative chemotherapy regimen (i.e. 1200 TBI or 200 TBI plus chemotherapy).
2. Previous treatment with Vemurafenib.
3. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
4. Systemic steroid therapy requirement.
5. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
7. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
8. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
9. History of coronary revascularization or ischemic symptoms.
10. Any patient known to have an LVEF less than or equal to 45 percent.
11. In patients > 60 years old, documented LVEF of less than or equal to 45 percent.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04-09; Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Determine the safety of the administration of vemurafenib in conjunction with ACT consisting of autologous TIL infused along with high dose aldesleukin following a non-myeloablative lymphodepleting preparative regimen. | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boni A, Cogdill AP, Dang P, Udayakumar D, Njauw CN, Sloss CM, Ferrone CR, Flaherty KT, Lawrence DP, Fisher DE, Tsao H, Wargo JA. Selective BRAFV600E inhibition enhances T-cell recognition of melanoma without affecting lymphocyte function. Cancer Res. 2010 Jul 1;70(13):5213-9. doi: 10.1158/0008-5472.CAN-10-0118. Epub 2010 Jun 15. PMID 20551059
- [Background] Dudley ME, Yang JC, Sherry R, Hughes MS, Royal R, Kammula U, Robbins PF, Huang J, Citrin DE, Leitman SF, Wunderlich J, Restifo NP, Thomasian A, Downey SG, Smith FO, Klapper J, Morton K, Laurencot C, White DE, Rosenberg SA. Adoptive cell therapy for patients with metastatic melanoma: evaluation of intensive myeloablative chemoradiation preparative regimens. J Clin Oncol. 2008 Nov 10;26(32):5233-9. doi: 10.1200/JCO.2008.16.5449. Epub 2008 Sep 22. PMID 18809613
- [Background] Chapman PB, Hauschild A, Robert C, Haanen JB, Ascierto P, Larkin J, Dummer R, Garbe C, Testori A, Maio M, Hogg D, Lorigan P, Lebbe C, Jouary T, Schadendorf D, Ribas A, O'Day SJ, Sosman JA, Kirkwood JM, Eggermont AM, Dreno B, Nolop K, Li J, Nelson B, Hou J, Lee RJ, Flaherty KT, McArthur GA; BRIM-3 Study Group. Improved survival with vemurafenib in melanoma with BRAF V600E mutation. N Engl J Med. 2011 Jun 30;364(26):2507-16. doi: 10.1056/NEJMoa1103782. Epub 2011 Jun 5. PMID 21639808